CLINICAL TRIAL: NCT03297203
Title: Role of Innate Lymphoid Cells in the Immunosuppression of Septic Shock
Brief Title: Innate Lymphoid Cells in Septic Shock
Acronym: CriSIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-24
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- groupe1 (Experimental): patients in septic shock (group 1) in the medical intensive care unit of the Timone Hospital.
  Interventions: Behavioral: Blood sample
- groupe 2 (Active Comparator): patients with a bacterial sepsis alone, during a 6 months period.
  Interventions: Behavioral: Blood sample

INTERVENTIONS:
Behavioral: Blood sample — The investigators will take two kits of blood samples for the group 1, one during the early stage of the septic shock (48 first hours of care) and one during the late stage of the disease (between the fourth and the sixth day). We'll take only one kit of blood samples for the group 2. One kit includes one EDTA tube (5 mL) and five Lithium Heparin tubes (25 mL). The immune mapping will be made by Julien Carvelli, a gold medalist resident, in the framework of a Master 2. The analyses will be made in the laboratory of immunology in the Conception Hospital (Pr Vivier's team).

SUMMARY:
Less than ten years after their intial description, the comprehension of Innate Lymphoid Cells (ILCs) biology is rapidly improving. They can be classified into four subgroups (ILCs 1, 2, 3 and NK cells) on the basis of their cytokine production and transcription factor expression.

They seem to be players in infectious diseases in animals but their role in human anti-bacterial defense remains unknown.

In this prospective work, the investigators will compare ILCs phenotyping in ICU patients managed for a septic shock, comparing them to ICU patients without any infectious disease on their inclusion. The investigators will also make a large immune mapping in all patients, to place ILCs in the global immune depressed state observed in septic patients.

DETAILED DESCRIPTION:
Septic shock is a major public health problem. Even if mortality is decreasing, it's still high. Sepsis is a heterogeneous syndrome that encompasses a gamut of immune responses occurring during the host's response to a serious, life-threatening infection. The immune phenotype in sepsis ranges from proinflammatory (systemic inflammatory response syndrome and cytokine storm syndrome) to anti-inflammatory (immune depressed state). In order to apprehend septic shock as a whole, investigators should made a whole immune mapping in each patient. Within immune mapping of septic shock patients, innate lymphoid cells (ILCs) have never been explored.

ILCs include natural killer (NK) cells and three other main subsets, ILC1, ILC2 and ILC3, referred as to 'helper-like ILCs'. Since their discovery, ILCs have been shown to contribute to wound healing and defense against infection, and studies have revealed critical aspects of their differentiation. They are studied by flow cytometry and much of the role of ILCs remains to be elucidated, especially in humans. Like T Helper cells, investigators think it could exist an imbalance of ILCs in the late course of septic shock which could participate to the immune depressed state and the increase of patients' mortality at this stage.

So, investigators want to realize a whole immune mapping in patients managed for a septic shock focusing particularly on the innate lymphoid cells. investigators think that ILC1s and ILC3s could be increased in the patients' blood in the early course of the disease and could participate to the cytokine storm syndrome. On the contrary, ILC2s could be increased in the late stage of the septic shock, in correlation with the immune suppressed state. investigators will compare the blood rates of ILCs in septic shock with the blood rates of ILCs in patients with a bacterial sepsis but without severity criteria.

investigators will include 30 patients in septic shock (group 1) in the medical intensive care unit of the Timone Hospital (RUM - Pr Gainnier) and 30 patients with a bacterial sepsis alone, during a 6 months period. investigatorswill take two kits of blood samples for the group 1, one during the early stage of the septic shock (48 first hours of care) and one during the late stage of the disease (between the fourth and the sixth day). investigators'll take only one kit of blood samples for the group 2. One kit includes one EDTA tube (5 mL) and five Lithium Heparin tubes (25 mL). The immune mapping will be made by Julien Carvelli, a gold medalist resident, in the framework of a Master 2. The analyses will be made in the laboratory of immunology in the Conception Hospital (Pr Vivier's team).

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* patient admitted to resuscitation for septic shock
* patient admitted to intensive care for a serious condition and with no progressive infection at the time of collection

Exclusion Criteria:

* Minor patient
* Patient with therepeutic limitations
* Bone marrow failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Secondary infections | 7 days
  Any secondary infection diagnosed in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud VANNESTE, Study Director — Assistance Publisque Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Carvelli J, Piperoglou C, Bourenne J, Farnarier C, Banzet N, Demerle C, Gainnier M, Vely F. Imbalance of Circulating Innate Lymphoid Cell Subpopulations in Patients With Septic Shock. Front Immunol. 2019 Sep 20;10:2179. doi: 10.3389/fimmu.2019.02179. eCollection 2019. PMID 31616411